CLINICAL TRIAL: NCT06052163
Title: Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Tolerability of Bumetanide in Patients With Alzheimer's Disease.
Brief Title: Bumetanide in Patients With Alzheimer's Disease
Acronym: BumxAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kyan Younes, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-69153
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Bumetanide

STUDY DESIGN:
Intervention Model Description: 1. Bumetanide low dose, 15 participants
  2. Bumetanide high dose, 15 participants
  3. Placebo, 10 participants
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bumetanide low dose (Active Comparator): 15 participants will take bumetanide low dose orally for 6 months and will be evaluated on cognitive and functional tests.
  Participants blood samples will be tested for levels of proteins involved in Alzheimer's disease.
  Interventions: Drug: Bumetanide
- Bumetanide high dose (Active Comparator): 15 participants will take bumetanide high dose orally for 6 months and will be evaluated on cognitive and functional tests.
  Participants blood samples will be tested for levels of proteins involved in Alzheimer's disease.
  Interventions: Drug: Bumetanide
- Placebo (Placebo Comparator): 10 participants will take placebo orally for 6 months and will be evaluated on cognitive and functional tests.
  Participants blood samples will be tested for levels of proteins involved in Alzheimer's disease.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bumetanide — Bumetanide is an FDA approved loop diuretic that has been used for more than three decades to treat edema, congestive heart failure, and hypertension across the life span. It has a well-known side effect profile. Most importantly it can cause dehydration and electrolyte imbalance especially at higher doses. This medication is given to individuals at the similar age group as Alzheimer's disease patients and Alzheimer's disease or cognitive impairment do not preclude its use in patients who need it for its FDA indications. At low doses and when titrated carefully, the medication is well tolerated. However, it has not been studied specifically in Alzheimer's disease patients.
  Other Names: Bumex
  Arms: Bumetanide high dose; Bumetanide low dose
Drug: Placebo — A placebo has no active properties and is taken orally.
  Arms: Placebo

SUMMARY:
This study aims to investigate bumetanide in patients with biologically confirmed Alzheimer's disease (AD). Bumetanide is a potent diuretic administered orally and is FDA approved for the treatment of edema and hypertension. Repurposing bumetanide as a medication for AD has been proposed based on data that demonstrated its ability to "flip" the APOE genotype-dependent transcriptomic signatures in AD mouse and cell culture models. Critically, this discovery was subsequently explored in Electronic Health Record cohorts, which revealed that among individuals over the age of 65, bumetanide exposure was significantly associated with a lower prevalence of AD in three independent datasets.

Primary Objective: To evaluate the safety and tolerability of bumetanide when administered to participants with biomarker-confirmed Alzheimer's disease.

Secondary Objective: To evaluate the clinical and biomarker effects of bumetanide in participants with mild cognitive impairment or mild dementia due to Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment or mild dementia due to Alzheimer's disease.
* Alzheimer's disease medications are planned to remain stable throughout.
* Willingness and ability to complete all aspects of the study including assessments, neuropsychological testing, and MRI.

Exclusion Criteria:

* Clinically significant abnormalities in screening laboratory tests
* Chronic liver disease
* Renal insufficiency
* Poorly managed hypertension
* Participants taking the following concomitant medications, based on the current Prescribing Information for bumetanide: lithium, drugs with ototoxic potential, drugs with nephrotoxic potential, probenecid, and indomethacin.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | 6 months
  Number of participants with adverse events including clinical signs and symptoms, change in vital signs, ECGs, laboratory safety tests, and suicidality assessments.

SECONDARY OUTCOMES:
Change from baseline in The Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog13) | 6 months
  The ADAS-Cog evaluates cognition and is scored from 0 to 90 points with a score of 0 indicating no impairment, and a score of 90 indicating maximum impairment
Changed from baseline in the clinical dementia rating scale sum of boxes (CDR-SoB) | 6 months
  CDR-SoB evaluates function with total possible score of 0 to 18 with higher scores indicating more impairment

CONTACTS AND LOCATIONS:
Overall Officials: Kyan Younes, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graber-Naidich A, Lee J, Younes K, Greicius MD, Le Guen Y, He Z. Bumetanide Exposure Association with Alzheimer's Disease Risk. Res Sq [Preprint]. 2023 Feb 28:rs.3.rs-2574215. doi: 10.21203/rs.3.rs-2574215/v1. PMID 36909637
- [Background] Taubes A, Nova P, Zalocusky KA, Kosti I, Bicak M, Zilberter MY, Hao Y, Yoon SY, Oskotsky T, Pineda S, Chen B, Jones EAA, Choudhary K, Grone B, Balestra ME, Chaudhry F, Paranjpe I, De Freitas J, Koutsodendris N, Chen N, Wang C, Chang W, An A, Glicksberg BS, Sirota M, Huang Y. Experimental and real-world evidence supporting the computational repurposing of bumetanide for APOE4-related Alzheimer's disease. Nat Aging. 2021 Oct;1(10):932-947. doi: 10.1038/s43587-021-00122-7. Epub 2021 Oct 11. PMID 36172600
- See also: Stanford Neurology & Neurological Sciences Clinical Trials — https://med.stanford.edu/neurology/research/clinicaltrials.html
- See also: Stanford Alzheimer's Disease Research Center Clinical Trials and Research Studies — https://med.stanford.edu/adrc/clinicaltrials.html